CLINICAL TRIAL: NCT03988114
Title: A Single-Arm, Global, Phase 4 Study of Abemaciclib, a CDK 4 & 6 Inhibitor, in Combination With Nonsteroidal Aromatase Inhibitors (Anastrozole or Letrozole) in Participants With Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Advanced Breast Cancer With Poor Prognostic Factors
Brief Title: A Study of Abemaciclib (LY2835219) in Participants With HR+, HER2- Advanced Breast Cancer
Acronym: proMONARCH
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategic decision due to emerging new data for patients with HR+, HER2- metastatic breast cancer.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17395; I3Y-MC-JPCX (Other: Eli Lilly and Company); 2019-001781-16 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib + NSAI (Experimental): Abemaciclib given orally and nonsteroidal aromatase inhibitor (NSAI) of physician's choice (anastrazole or letrozole) given orally.
  Interventions: Drug: Abemaciclib; Drug: Nonsteroidal Aromatase Inhibitor (NSAI)

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Nonsteroidal Aromatase Inhibitor (NSAI) — Letrozole administered orally or anastrozole administered orally (physician choice)

SUMMARY:
The reason for this study is to see if the drug abemaciclib in combination with nonsteroidal aromatase inhibitors (anastrozole or letrozole) is effective in participants with Hormone Receptor Positive (HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) advanced breast cancer that have certain disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed (neo) adjuvant endocrine therapy and have cancer return after at least 12 months or have de novo cancer that has spread to other organs at diagnosis
* Participants must have 1 or more of the following:

  * A high grade tumor in tissue
  * Negative progesterone receptor (PR) status
  * Have cancer that has spread to the liver
  * Have a treatment-free interval (TFI) <36 months
* Participants must have HR+, HER2- breast cancer
* Participants must have adequate organ function

Exclusion Criteria:

* Participants must not have cancer that has spread to other organs that has severely affected their function
* Participants must not have cancer that has spread to the brain that is unstable or untreated
* Participants must not have received endocrine therapy in the metastatic setting
* Participants must not have known active infection
* Participants must not have received prior endocrine therapy and had disease return within 12 months from completion of treatment
* Participants must not have received prior treatment with any cyclin-dependent kinase (CDK) 4 & 6 inhibitor or everolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-16 (Estimated); Primary Completion 2022-03-23 (Estimated); Study Completion 2023-03-23 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Baseline to Progressive Disease or Death from Any Cause (Estimated up to 26 Months)
  PFS
Objective Response Rate (ORR): Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) | Baseline to Objective Disease Progression (Estimated up to 26 Months)
  ORR

SECONDARY OUTCOMES:
Duration of Response (DoR) | Date of CR or PR to Date of Objective Disease Progression or Death from Any Cause (Estimated up to 26 Months)
  DoR
Disease Control Rate (DCR): Percentage of Participants with a Best Overall Response of CR, PR, or Stable Disease (SD) | Baseline to Objective Disease Progression (Estimated up to 26 Months)
  DCR
Clinical Benefit Rate (CBR): Proportion of Participants with Best Overall Response of CR, PR, or SD with Duration of SD for at Least 6 Months | Date of CR, PR or SD to 6 Months Post CR, PR or SD (Estimated up to 26 Months)
  CBR
Time to Response (TTR) | Baseline to Date of CR or PR (Estimated up to 26 Months)
  TTR

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (119):
- United States (70):
  - Southern Cancer Center, P.C., Daphne, Alabama
  - Arizona Oncology Associates, P.C., Tempe, Arizona
  - Compassionate Cancer Care Medical Group Inc, Fountain Valley, California
  - California Cancer Associates Research and Excellence (cCARE), Fresno, California
  - Beaver Medical Group, Highland, California
  - Pacific Cancer Care, Monterey, California
  - St. Joseph Hospital, Orange, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - California Cancer Associates in Research and Excellence, San Marcos, California
  - Cancer Center of Santa Barbara with Sansum Clinic, Santa Barbara, California
  - UCLA Medical Center, Torrance, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center, Lone Tree, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - BayCare Medical Group, Clearwater, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Cancer Specialists of North Florida -St Augustine, Saint Augustine, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Cleveland Clinic of Florida, Weston, Florida
  - Summit Cancer Care, Savannah, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Central Maine Medical Center, Lewiston, Maine
  - York Hospital, York Village, Maine
  - HCA Midwest, Kansas City, Missouri
  - Oncology Hematology West, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Valley Health System, Paramus, New Jersey
  - Broome Oncology LLC, Johnson City, New York
  - Abington Hematology Oncology Associates, Horsham, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Oncology - Abilene, Abilene, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology P.A., Dallas, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Marnie McFadden Ward Cancer Center, Dallas, Texas
  - Texas Oncology P.A., El Paso, Texas
  - Texas Oncology Flower Mound, Flower Mound, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Renovatio Clinical, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Texas Oncology- Mesquite, Mesquite, Texas
  - Texas Oncology - Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology - Paris, Paris, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - US Oncology, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology-Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology-Wichital Falls Texoma Cancer Center, Wichita Falls, Texas
  - Intermountain Medical Center, St. George, Utah
  - Hematology Oncology Associates of Fredericksburg Inc., Fredericksburg, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Salem, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
- Argentina (8):
  - Centro de Oncologia e Investigacion Buenos Aires, Berazategui, Buenos Aires
  - CEMEDIC, CABA, Buenos Aires
  - CENIT Centro de Neurociencias, Investigación y Tratamiento, CABA, Ciudad Autonoma Buenos Aires
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Clinica Adventista de Belgrano, Ciudad Autonoma Buenos Aires
  - Sanatorio Parque, Salta
  - Centro Polivalente de Asistencia e Inv. Clinica CER-San Juan, San Juan
  - Centro para la Atencion Integral del Paciente Oncologico, Tucumain
- Austria (4):
  - Universitätsklinikum Graz, Graz, Styria
  - Universitätsklinik Innsbruck, Innsbruck, Tyrol
  - Universitätsklinikum Salzburg, Salzburg
  - AKH, Vienna
- Belgium (4):
  - Algemeen Ziekenhuis St Jan Brugge, Bruges
  - Hopital De Jolimont, Haine-St.- Paul
  - VZW REgional Ziekenhuis Jan Yperman, Ieper
  - Clinique Saint Pierre Ottignies, Ottignies
- Brazil (15):
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Instituto de Cancer de Londrina, Londrina, Paraná
  - Instituto COI de Pesquisa Educação e Gestão, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade Ijui, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born de Lajeado, Lajeado, Rio Grande do Sul
  - Hospital São Lucas - PUCRS - ONCOLOGY, Porto Alegre, Rio Grande do Sul
  - Fundação PIO XII, Barretos, São Paulo
  - Hospital das Clinicas da FMRP, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital de Base Fac de Medicina de Sao Jose do Rio Preto, Sao Jose Rio Preto, São Paulo
  - INCA - Instituto Nacional Do Cancer, Rio de Janeiro
  - Soc. Beneficente de Senhoras Hospital Sirio Libanes-Oncology, São Paulo
  - Clin. Pesq.e Centro Estudos Oncologia Ginecológica e Mamária, São Paulo
  - Fundacao Antonio Prudente-Hosp. do Cancer AC Camargo, São Paulo
  - Clinica Onco Star, São Paulo
- Germany (3):
  - Hämatologisch-Onkologische Praxis Augsburg, Augsburg, Bavaria
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - St. Vincenz-Krankenhaus GmbH-Frauen- und Kinderklinik St. Louise, Paderborn
- Italy (7):
  - Istituto Tumori Fondazione G. Pascale IRCCS, Napoli, Naples
  - Fondazione Piemonte l'Oncologia-Istituto Ricerca Cura Cancro, Candiolo, Torino
  - Policlinico S. Orsola Malpighi - Universita di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Ospedale San Martino di Genova, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto, Padua
  - Centro di Riferimento Oncologico, Udine
- Puerto Rico (2):
  - Puerto Rico Hematology/Oncology Group, Bayamón, PR
  - Ad-Vance Medical Research, Ponce
- Taiwan (6):
  - E-DA Cancer Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - Koo Foundation Sun Yan-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) in Participants With HR+, HER2- Advanced Breast Cancer — https://www.lillytrialguide.com/en-US/studies/metastatic-breast-cancer/JPCX